CLINICAL TRIAL: NCT04601974
Title: Phase I/IIa, First-in-human, Open-label, Single-site Trial of In-vivo Lentiviral Engineered Potassium (K+) Channel (EKC) Gene Therapy for Refractory Epilepsy
Brief Title: Lentiviral Gene Therapy for Epilepsy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/0202
Record Dates: First submitted 2020-10-06; First posted 2020-10-26 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Drug Resistant Epilepsy
Keywords: lentiviral gene therapy; brain; surgery; drug resistant epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lentiviral gene therapy treatment (Intervention Arm) (Experimental): Patients will receive a single dose of lentiviral gene therapy treatment administered once intracranially
  Interventions: Genetic: lentiviral gene therapy

INTERVENTIONS:
Genetic: lentiviral gene therapy — lentiviral gene therapy to treat drug resistant epilepsy

SUMMARY:
This is a phase I/IIa clinical trial investigating the safety of a lentiviral epilepsy gene therapy using an engineered potassium channel in patients with refractory epilepsy.

DETAILED DESCRIPTION:
Epilepsy affects about 1% of the population. One third of affected individuals continue to have seizures despite optimal medication. The only realistic prospect of seizure freedom, feasible in very few cases, is surgery to remove the brain area where seizures arise.

Patients with refractory neocortical epilepsy who are being evaluated for surgical resection of the seizure focus will be invited to join the trial. The non-integrating lentiviral vector, which has been engineered to deliver an engineered potassium channel, will be administered via intracerebral infusion to the area scheduled for resection.

The primary objective in this study is to test the safety of the lentiviral gene therapy treatment, including the surgical procedures required for vector administration. Secondary objectives will look at delayed onset adverse events and indicators of efficacy.

ELIGIBILITY:
Inclusion Criteria:

SCREENING/PRE-CONSENT:

1. Female and male patients with refractory focal epilepsy
2. Aged ≥ 18 years (no upper age limit but deemed medically fit for surgery with a life expectancy of at least 5 years)
3. Patient lives within 1 hour of transfer to an acute neurosurgical unit
4. Being considered for resective brain surgery (to remove the epileptogenic focus) based on first-stage preoperative assessments carried out as part of routine clinical care within 2 years of registration, showing:

   4.1. Absence of vascular brain lesions or vascular malformations and/or cancer in the resection area (as confirmed on MRI) 4.2. Absence of active, untreated psychiatric disease in the opinion of the treating clinician (as confirmed by neuropsychiatric assessment) 4.3. Patient requires second-stage intracranial EEG investigations to be carried out via burr hole surgery to further assess eligibility for resective brain surgery

   PRE-REGISTRATION:
5. Patient deemed clinically suitable for resective brain surgery (i.e. a single region of seizure onset in the neocortex has been identified, and it does not overlap with areas necessary for critical functions such as language), as confirmed by intracranial EEG investigations
6. Patients who are women of childbearing potential (WOCBP), or male patients with female partners who are WOCBP or pregnant must agree to use highly effective methods of contraception from the time consent is signed until three months after treatment. Men (if applicable), must also advise their female partners regarding contraceptive requirements as listed for female patients who are WOCBP or pregnant.
7. Able and willing to give written informed consent to join trial

Exclusion Criteria:

1. Not deemed clinically suitable for resective brain surgery (e.g. because of failure to identify a single region of seizure onset in the neocortex, region is too extensive or the region overlaps with areas necessary for critical functions such as language), as confirmed by intracranial EEG investigations
2. Vascular brain lesions or vascular malformations in area of planned resection
3. Detection of active cancer or on systemic treatment for cancer
4. Known or suspected HIV infection (confirmed by PCR test) and/or taking antiretroviral therapy
5. Patient deemed medically unfit for anaesthesia and surgery
6. Active, untreated psychiatric disease in the opinion of the treating clinician
7. Concurrent and/or recent involvement in another clinical trial of an investigational medicinal product (within last 3 months)
8. Females who are pregnant (confirmed by serum/urine ß-HCG) or actively breast-feeding
9. Known allergies to excipients of lentiviral gene therapy
10. Patient unlikely to cooperate with a 5-year follow-up; medical or psychological condition at the discretion of the investigator which would not permit compliance with the protocol or meaningful written informed consent
11. Any other known condition which is assessed as an intolerable risk by the investigator upon inclusion in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Safety during the First Year (for adverse events related to lentiviral gene therapy only) | At 6 weeks, 3 months, 6 months and 12 months after trial treatment
  Number and severity of all adverse events (graded using CTCAE v5.0) in patients deemed causally related to lentiviral gene therapy
Safety during the First Year (for adverse events causally related to investigational surgical procedures only) | At 6 weeks, 3 months, 6 months and 12 months after trial treatment
  Number and severity of all adverse events (graded using CTCAE v5.0) deemed causally related to any of the investigational surgical trial procedures required for vector administration

SECONDARY OUTCOMES:
Long-Term Safety (for adverse events related to lentiviral gene therapy only) | From 1 to 5 years after treatment
  Number of serious adverse events (graded using CTCAE v5.0) in patients related to the lentiviral gene therapy
Long-Term Safety (for adverse events causally related to investigational surgical procedures only) | From 1 to 5 years after treatment
  Number of serious adverse events (graded using CTCAE v5.0) in patients related to the investigational surgical procedures required for vector administration
Clinical Indicators of Efficacy and Tolerability | Measured at 6 weeks, 3 months, 6 months, and 12 months/1 year after trial treatment
  Seizure frequency and severity over preceeding 4 weeks
Clinical Indicators of Efficacy and Tolerability | Measured at 12 months/1 year, 2 years, 3 years, 4 years and 5 years after trial treatment
  Seizure frequency and severity (using IALE outcomes scale)
Clinical Indicators of Efficacy and Tolerability | at 3, 6, or 12 months, or at 2, 3, 4, and 5 years after trial treatment
  Proportion of patients who have had surgical resection
Cortical excitability | at 6 months after trial treatment (only for patients in TMS study)
  Cortical excitability (assessed using TMS, EMG, and high-density EEG)

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared with other researchers who are working in the public and charitable sector (universities, research institutes) or commercial companies involved in health care research in the UK or overseas. Participant data will be fully anonymised prior to data sharing. This means there will be no way to link the data to the original data set, or to individual participants. Anonymisation will be done by the trial statistician. Data shared in this way will be protected by a contractual agreement put in place between UCL (the Sponsor) and any respective institution.